CLINICAL TRIAL: NCT03755843
Title: PREDICTION OF FLUID RESPONSIVENESS WITH PASSIVE LEG RISING IN PREGNANT PATIENTS WITH SEVERE PREECLAMPSIA
Status: Completed | Type: Observational
Sponsor: RAUL CARRILLO ESPER (Other)
Responsible Party: Sponsor-Investigator, RAUL CARRILLO ESPER, GMEMI coordinator, Grupo Mexicano para el Estudio de la Medicina Intensiva
Organization: Grupo Mexicano para el Estudio de la Medicina Intensiva (Other)
Other Study IDs: DI/17/112/03/039
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Pre-Eclampsia; Volume Overload; Hemodynamic Instability
Keywords: passive leg risging; Fluid challenge; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PASSIVE LEG RISING — Pasive Leg Rising: In the supine method, the legs are lifted passively from the horizontal position to a 30° to 45° elevation while the head of the bed is flat.
  Fluid Challenge: Fluid responsiveness is generally defined as an increase in SV or CO of 10% to 15% in response to a 250 mL crystalloid fluid bolus
  Other Names: fluid challenge

SUMMARY:
BACKGROUND: A cornerstone of treatment in preeclampsia is to correct the potential hypovolemia with intravascular optimisation, which is usually performed as a fluid challenge. The prediction of fluid responsiveness in these patients, secondary to anatomical and physiological changes associated with pregnancy has not been established. This study aims to evaluate if Passive Leg Raising (PLR) protocol can predict fluid responsiveness in pregnant patients with severe preeclampsia.

MATERIALS AND METHODS: in 35 pregnant women diagnosed with preeclampsia with a clinical indication to optimise intravascular volume, . A PLR manoeuvre and a fluid challenge will be performed, and hemodynamic parameters were recorded using Bioreactance technology. Descriptive statistical analyses, Pearson chi-square test, and mean standard deviation (SD) will be calculated. Analysis of proportion was used to calculate probabilistic intersections of the interventions. The area under curve, sensitivity, specificity, positive predictive value and negative predictive value were calculated for a delta of 12.

Objective: to evaluate the if passive leg rising protocol identifies fluid responsivness in pregnant patients with preeclampsia

DETAILED DESCRIPTION:
INTRODUCTION The clinical manifestations of preeclampsia (PE) are the consequence of endothelial dysfunction. [1, 2] Different hemodynamic patterns have been described, which includes: high vascular resistance, cardiac output (CO) alterations, relative hypovolemia, and increased risk for pulmonary oedema, [3-6] which has been recognised as the most common final cause of death in women with complications of hypertension7. The risk of pulmonary oedema in preeclampsia is caused by different pathophysiological changes that follow the disease. It can be classified as increase preload caused by iatrogenic resuscitation and resolving puerperal oedema. Cardiac causes such as the presence of a myopathic ventricle, diastolic dysfunction, valvular heart disease, increased afterload caused by severe hypertension and increased vascular resistance, and other factors such as reduced oncotic pressure increased capillary permeability or a combination of all.

A cornerstone of treatment to correct the potential hypovolemia in preeclampsia is intravascular volume optimization, which usually is performed as a fluid challenge, [8-9] However, the increased risk of pulmonary oedema has made us understand the need to use dynamic hemodynamic parameters for fluid responsiveness to guide optimal intravascular volume optimization in this group of patients.

Monitoring fluid therapy upon clinical observation or the estimation of filling pressures using clinical markers such as blood pressure, pulse rate and urinary output as an endpoint of euvolemia may be inaccurate in women with severe preeclampsia. In critically ill settings the resolution of severe hypovolaemia is accompanied by rising blood pressure, falling of pulse rate and increasing the urinary output. However, in preeclamptic women, oliguria may develop because of intrinsic renal disease and may not respond to plasma volume expansion with an increase of urinary output. [20] Tachycardia commonly complicates severe preeclampsia, and a persistently rapid pulse rate may not be a reliable indication of intravascular volume depletion, especially when the systolic blood pressure is within reasonable limits.

In the intensive care unit, patients with spontaneous ventilation, an increase of stroke volume during passive leg raising (PLR) predicts fluid responsiveness. [10-13] However, during pregnancy, the validity of PLR has been questioned, secondary to the known anatomical changes that occur from the compression of the inferior vena cava (IVC) by the gravid uterus and the presence of increased abdominal pressure. [14-16] However recently Brun20 published the first study that showed that PLR accurately predicts fluid responsiveness in the setting of Severe Preeclampsia.

Thoracic bioreactance technology, [17] which is based on the analysis of thoracic voltage amplitude changes in response to a high-frequency injected current, and has the potential to be a useful noninvasive clinical tool for monitoring hemodynamics in pregnant women. However, the prediction of fluid responsiveness in these patients, secondary to anatomical and physiological changes associated with pregnancy has not been established.

The objective of this protocol is to evaluate if PLR test can predict fluid responsiveness in pregnant patients with severe preeclampsia.

MATERIALS AND METHODS The study is approved by the Institutional Review Board. Both ethic and research committee approved the protocol with registers number DI/17/112/03/039. Patients will be informed and signed consent before participation. Patients are going to be prospectively assessed, and consecutive measurements will be performed in an obstetric ICU of Mexico´s General Hospital Dr Eduardo Liceaga from December 2016 to July 2017. A sample was calculated for known variance P .01. Measurements for blood pressure and heart rate are made using bioreactance (NICOMTM Panamedical Mexico City, Mexico) technology.[18] The monitor will be placed at bedside, to monitor Systolic Arterial Pressure (SAP) and Diastolic Arterial Pressure (DAP), Stroke Volume (SV), Stroke Volume Index (IVS), Cardiac Output (CO) and Cardiac Index (CI).18 Because hemodynamic values may vary within a respiratory cycle,[17] an average of 10 consecutive cardiac cycles, over at least one respiratory cycle, was used for measurements of SAP, DAP, MAP, SV, and ISV.

Moreover, we use the best dynamic index report under those 10 minutes. A PLR manoeuvre was performed for 3 minutes. The manoeuvre involved elevating the patient's legs and placing them on an inflatable leg wedge providing an angle of 45 degrees while in the supine position. Next, a 250 crystalloid /colloid (Hartmann + albumin 25%) bolus was given recording the same hemodynamic parameters to observe changes in dynamic measurements to compare both results and classified them as responder and non-responder. No determination or Central Venous Pressure or surrogate was made because of the accumulative evidence of the failure of this methods to detect changes in intravascular volume status. A change of 12% after PLR and bolus was used to consider a patient responder[20]. Finally, we used the values for ISV because it would be the better parameter (without the influence of heart rate and independent of the body area).

STATISTICAL ANALYSIS Using SPSS 23 statistics Descriptive data analysis of patients will be performed for this purpose, a multivariable database will be constructed, and descriptive statistical analyses made. To evaluate the distribution between variables a Pearson chi-square test will be used. Mean standard deviation (SD) values, and analysis of proportion with the aim of knowing the probabilistic intersections. The area under the curve, sensitivity, specificity, negative predictive and positive predictive value will be calculated for 12 for ISV.

ELIGIBILITY:
Inclusion Criteria:

second and thrith trimestrer Pregnant women with severe preeclampsia Non intubated

Exclusion Criteria:

Amputation of any limb heart or valve disease Chronic renal failure Chronic Liver failure

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — second a thirth pregnant women
Study Population: Female pregnant women with sever preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Passive Leg Rising | 6 months
  evaluate if PLR test can predict fluid responsiveness in pregnant patients with severe

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Mexico, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duley L. The global impact of pre-eclampsia and eclampsia. Semin Perinatol. 2009 Jun;33(3):130-7. doi: 10.1053/j.semperi.2009.02.010. PMID 19464502
- [Background] Sibai B, Dekker G, Kupferminc M. Pre-eclampsia. Lancet. 2005 Feb 26-Mar 4;365(9461):785-99. doi: 10.1016/S0140-6736(05)17987-2. PMID 15733721
- [Background] Young P, Johanson R. Haemodynamic, invasive and echocardiographic monitoring in the hypertensive parturient. Best Pract Res Clin Obstet Gynaecol. 2001 Aug;15(4):605-22. doi: 10.1053/beog.2001.0203. PMID 11478818
- [Background] Barton JR, Sibai BM. Life-threatening emergencies in preeclampsia-eclampsia. J Ky Med Assoc. 2006 Sep;104(9):410-8. No abstract available. PMID 17100119
- [Background] Sciscione AC, Ivester T, Largoza M, Manley J, Shlossman P, Colmorgen GH. Acute pulmonary edema in pregnancy. Obstet Gynecol. 2003 Mar;101(3):511-5. doi: 10.1016/s0029-7844(02)02733-3. PMID 12636955
- [Background] Societe francaise d'anesthesie et de reanimation (Sfar); College national des gynecologues et obstetriciens francais (CNGOF); Societe francaise de medecine perinatale (SFMP); Societe francaise de neonatalogie (SFNN). [Multidisciplinary management of severe pre-eclampsia (PE). Experts' guidelines 2008. Societe francaise d'anesthesie et de reanimation. College national des gynecologues et obstetriciens francais. Societe francaise de medecine perinatale. Societe francaise de neonatalogie]. Ann Fr Anesth Reanim. 2009 Mar;28(3):275-81. doi: 10.1016/j.annfar.2009.02.015. Epub 2009 Mar 24. No abstract available. French. PMID 19321292
- [Background] Sibai BM, Mabie BC, Harvey CJ, Gonzalez AR. Pulmonary edema in severe preeclampsia-eclampsia: analysis of thirty-seven consecutive cases. Am J Obstet Gynecol. 1987 May;156(5):1174-9. doi: 10.1016/0002-9378(87)90135-9. PMID 3578433
- [Result] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Result] Monnet X, Teboul JL. Passive leg raising. Intensive Care Med. 2008 Apr;34(4):659-63. doi: 10.1007/s00134-008-0994-y. Epub 2008 Jan 23. PMID 18214429
- [Result] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963
- [Result] Brun C, Zieleskiewicz L, Textoris J, Muller L, Bellefleur JP, Antonini F, Tourret M, Ortega D, Vellin A, Lefrant JY, Boubli L, Bretelle F, Martin C, Leone M. Prediction of fluid responsiveness in severe preeclamptic patients with oliguria. Intensive Care Med. 2013 Apr;39(4):593-600. doi: 10.1007/s00134-012-2770-2. Epub 2012 Dec 6. PMID 23223774
- [Result] Vartun A, Flo K, Acharya G. Effect of passive leg raising on systemic hemodynamics of pregnant women: a dynamic assessment of maternal cardiovascular function at 22-24 weeks of gestation. PLoS One. 2014 Apr 14;9(4):e94629. doi: 10.1371/journal.pone.0094629. eCollection 2014. PMID 24732308
- [Result] Marques NR, Martinello C, Kramer GC, Costantine MM, Vadhera RB, Saade GR, Hankins GD, Pacheco LD. Passive leg raising during pregnancy. Am J Perinatol. 2015 Mar;32(4):393-8. doi: 10.1055/s-0034-1389089. Epub 2014 Sep 21. PMID 25241109